CLINICAL TRIAL: NCT07333092
Title: Investigation of the Effects of Proprioceptive Exercises on Balance, Kinesiophobia, and Functionality After Anterior Cruciate Ligament Surgery: A Randomized Controlled Trial
Brief Title: Investigation of the Effects of Proprioceptive Exercises After Anterior Cruciate Ligament Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Assoc.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar80
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): balance exercises
  Interventions: Other: control
- exercise group (Experimental): balance exercises + proprioceptive exercises
  Interventions: Other: control; Other: exercise

INTERVENTIONS:
Other: control — Patients will only be given balance exercises that are currently available at the hospital.
Other: exercise — In addition to balance exercises, proprioceptive exercises will be performed.
  Arms: exercise group

SUMMARY:
The aim of this study is to investigate the effects of proprioceptive exercises on balance, kinesiophobia, and functionality after anterior cruciate ligament surgery.

DETAILED DESCRIPTION:
A sociodemographic form will be used to obtain sociodemographic information, the y-balance test will be used to assess balance at the beginning and end of the study, the Tampa Kinesiophobia Scale will be used to assess kinesiophobia, and the Lysholm Knee Score Scale will be used to assess functionality. Both groups will perform balance exercises currently offered at the hospital. The experimental group will also receive proprioceptive exercises in addition to the balance exercises currently offered at the hospital. The exercises will be performed three days a week for 12 weeks for both groups. In this study, the independent variables are the addition or non-addition of proprioceptive exercises, while balance, kinesiophobia, and functionality are the dependent variables. The significance levels of the obtained data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria

* Being between 20-40 years of age
* Having undergone anterior cruciate ligament (ACL) surgery
* Being in the 2nd week of rehabilitation after ACL surgery

Exclusion Criteria

* Having a concomitant meniscus injury
* Having a concomitant medial collateral ligament injury
* Being in the 1st week of rehabilitation after ACL surgery

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Lysholm Knee Scoring Scale | 14 weeks
  The Lysholm scale was developed for use by physicians and has been verified in patients with Anterior Cruciate Ligament and meniscal injuries. It's also been approved as a patient-administered tool for assessing symptoms and function in people who have had a variety of knee injuries. The Lysholm scale assesses the domains of symptoms and complaints, as well as functioning in daily activities, however, it doesn't assess the area of sports and recreational activities. There are 8 items on this questionnaire and graded on a scale of 0 to 100, with higher scores suggesting fewer symptoms and better function
Tampa Kinesiophobia Questionnaire | 14 weeks
  Tampa Kinesiophobia Questionnaire is a 17-question questionnaire that assesses avoidance of injury and fear of movement. The scale is scored using a Likert scale (1 = Strongly disagree, 4 = Strongly agree). Items 4, 8, 12 and 16 are reversed to calculate the total score of the scale. The total score is between 17 and 68. As the score of the person increases, it is understood that their kinesiophobia is high. A total score higher than 37 is considered as high kinesiophobia. However, since not every item of the questionnaire addresses patients with headache in this study, some questions were removed, some questions were edited and some questions were added to create a kinesiophobia questionnaire for headache. The newly created questionnaire consists of 23 items. Again, it is scored using a Likert scale with "1 = Strongly disagree, 4 = Strongly agree". As the score increases, it is understood that the level of kinesiophobia is high
Y Balance Test | 14 weeks
  The Y Balance Test will be used to assess dynamic balance by measuring reach distances in three directions (anterior, posteromedial, and posterolateral) while standing on one leg. Each direction will be tested three times, and the average reach distance will be normalized to leg length. A composite score will be calculated and expressed as a percentage to evaluate overall dynamic balance capacity. Higher scores indicate better balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe ŞAN, Study Chair — Uskudar University
Locations (1):
- Şanlıurfa Mehmet Akif İnan Health Application and Research Center, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zult T, Gokeler A, van Raay JJAM, Brouwer RW, Zijdewind I, Farthing JP, Hortobagyi T. Cross-education does not accelerate the rehabilitation of neuromuscular functions after ACL reconstruction: a randomized controlled clinical trial. Eur J Appl Physiol. 2018 Aug;118(8):1609-1623. doi: 10.1007/s00421-018-3892-1. Epub 2018 May 23. PMID 29796857
- [Background] Erayata BN, Menek B. Investigating the effects of percussion massage therapy on pain, functionality, muscle diameter, and proprioception in individuals with ACL reconstruction: a randomized controlled trial. PLoS One. 2025 Mar 26;20(3):e0319731. doi: 10.1371/journal.pone.0319731. eCollection 2025. PMID 40138389
- [Background] Keays SL, Bullock-Saxton JE, Newcombe P, Bullock MI. The effectiveness of a pre-operative home-based physiotherapy programme for chronic anterior cruciate ligament deficiency. Physiother Res Int. 2006 Dec;11(4):204-18. doi: 10.1002/pri.341. PMID 17236528